CLINICAL TRIAL: NCT03584802
Title: Therapeutic Plasma Exchange, Rituximab and Intravenous Immunoglobulins for Severe Acute Exacerbation of Idiopathic Pulmonary Fibrosis Admitted in ICU: an Open, Randomized, Controlled Trial
Brief Title: Therapeutic Plasma Exchange, Rituximab and IV Ig for Severe Acute Exacerbation of IPF Admitted in ICU
Acronym: EXCHANGE-IPF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P160915J
Record Dates: First submitted 2018-06-06; First posted 2018-07-12 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Exacerbation of Idiopathic Pulmonary Fibrosis
Keywords: severe acute exacerbation of idiopathic pulmonary fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental treatment of AE-IPF (Experimental): The experimental group will receive a combination of: 1- Methylprednisolone bolus of 1g IV day 1, then 20 mg/day (or oral prednisolone equivalent) for 21 days; 2- Nine therapeutic plasma exchanges of 1,5x the estimated plasma volumes using albumin: saline (3:1) or fresh frozen plasma in case of an INR superior to 1,5, on days 1,2,3,5,7,9,11,13,15; followed by administration of low dose of intravenous immunoglobulin (100mg/kg) 3, Rituximab 1g IV on days 7 and 15 (after therapeutic plasma exchange and premedication) 4, Intravenous immunoglobulin 0,5g/kg/d on days 16 to 19,
  Interventions: Other: Therapeutic plasma exchanges
- Conventional treatment of AE-IPF (Active Comparator): Intravenous methylprednisolone bolus of 10mg/kg on day1, 2 and 3, then 1mg/kg/d for 1 week, and 0,75 mg/kg/d for 1 week, then 0,5 mg/kg/d for 1 week, and 0,25 mg/kg/d for 1 week, and 0,125 mg/kg/d until day 90. Shift to oral prednisone as soon as the oral route is available.
  Interventions: Other: Conventional treatment of AE-IPF

INTERVENTIONS:
Other: Therapeutic plasma exchanges — The patient will initially receive Methylprednisolone bolus of 1g i.v. day 1, then 20 mg/day (or oral prednisone equivalent) for 21 days; and then he will have nine therapeutic plasma exchanges of 1.5x the estimated plasma volumes using albumin:saline (3:1) or fresh frozen plasma in case of an INR superior to 1.5, on days 1,2,3,5,7,9,11,13,15; followed by administration of low dose of intravenous immunoglobulin (100 mg/kg). On days 7 and 15, the patient will receive rituximab 1 g i.v. on days 7 and 15 (after therapeutic plasma exchange and premedication); and intravenous immunoglobulin 0.5 g/kg/d on days 16 to 19.
  Arms: Experimental treatment of AE-IPF
Other: Conventional treatment of AE-IPF — Conventional treatment of AE-IPF
  Arms: Conventional treatment of AE-IPF

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a fibroproliferative, irreversible disease of unknown cause, occurring mainly in patients older than 50. IPF is a rare but fatal lung disease, with an estimated prevalence of 14 to 28/100000 and a median survival time of 3 years. Acute exacerbation of IPF (AE-IPF) is a major event of IPF, as it is responsible for the death of 30-50 % of IPF patients; its annual incidence varies between 5 and 10%. The current literature indicates that IPF is associated with the development of an auto-immunity process targeting epithelial and endothelial lung cells. Autoantibodies have been associated with a poorer prognosis. A study by DONAHOE et al. (Plos One, 2015) indicates that the combination of corticosteroids, plasma exchanges, rituximab and immunoglobulins may improve the prognosis of the most severe forms of AE-IPF. In that study, the observed survival rate in patients receiving this combination of treatment was 70% as compared with 20% in historical controls. This therapeutic combination approach is designed both to eliminate and inhibit the production of circulating antibodies targeting the lungs. Considering the high mortality rate of an AE-IPF episode and the potential benefit of such an original approach, a well-conducted randomized controlled trial is critical.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis (IPF) is a fibroproliferative, irreversible disease of unknown cause, occurring mainly in patients older than 50. IPF is a rare but fatal lung disease, with an estimated prevalence of 14 to 28/100000 and a median survival time of 3 years. Acute exacerbation of IPF (AE-IPF) is a major event of IPF, as it is responsible for the death of 30-50 % of IPF patients; its annual incidence varies between 5 and 10%. The current literature indicates that IPF is associated with the development of an auto-immunity process targeting epithelial and endothelial lung cells. Autoantibodies have been associated with a poorer prognosis. A study by DONAHOE et al. (Plos One, 2015) indicates that the combination of corticosteroids, plasma exchanges, rituximab and immunoglobulins may improve the prognosis of the most severe forms of AE-IPF. In that study, the observed survival rate in patients receiving this combination of treatment was 70% as compared with 20% in historical controls. This therapeutic combination approach is designed both to eliminate and inhibit the production of circulating antibodies targeting the lungs. Considering the high mortality rate of an AE-IPF episode and the potential benefit of such an original approach, a well-conducted randomized controlled trial is critical.

The main objective is to evaluate the impact on overall mortality at day 28 of plasma exchanges, rituximab, intravenous immunoglobulins (IVIg), and corticosteroid administration versus standard corticosteroid therapy in hypoxemic patients admitted in ICU for severe acute exacerbation of idiopathic pulmonary fibrosis.

The primary assessment criterion will be overall mortality at day 28 after initiation of therapy (Day 1).

Secondary objectives are the following:

1. Efficacy:

   1.1. To compare the overall mortality at day 90, at 6 months and at 12 months after the initiation of therapy 1.2. To compare the exposition to mechanical ventilation 1.3. To compare the length of ICU and hospital-stay 1.4. To compare the evolution of Sequential Organ Failure Assessment (SOFA) score 1.5. To compare the radiological evolution 1.6. To compare the evolution of lung injury biomarkers in plasma 1.7. To compare the changes in circulating autoantibodies levels before and after therapy 1.8. To compare the evolution of blood fibrocytes proportion 1.9. To evaluate respiratory functional at 3 months and compare data previously available.

   1.10. To assess quality of life (SF36), autonomy (ADL) and muscle strength scores (MRC) at 3 months of inclusion (Cf annexe)
2. Safety:

   2.1. To compare the occurrence of healthcare-associated infection 2.2. To describe the specific complications associated to the experimental treatment

   Secondary assessment criteria are the following:
3. Efficacy:

   3.1. Overall mortality at day 90, at 6 months and at 12 months 3.2. Number of days alive without mechanical ventilation between inclusion and day 28 3.3. Length of ICU-stay and hospital-stay 3.4. Changes in SOFA score from D1 to D3, D7, D16, D21, D28 or discharge-day from ICU as appropriate 3.5. Variation of global extent of High Resolution Computed Tomography (HRCT) infiltrates between initial HRCT and D90 3.6. Changes in lung injury plasmatic biomarkers (KL-6, SP-D) from D1 to D16, D21, D28 and D90 3.7. Changes in circulating antibodies levels (anti-periplakin, anti-HSP70 and anti-vimentin antibodies) from D1 to D28 and D90 3.8. Changes in the proportion of blood fibrocytes from D1 to D16, D28 and D90
4. Safety:

4.1. Proportion of patients with at least one episode of any healthcare-associated infection between inclusion and D28 4.2. The following complications in the experimental group will be described: 4.2.1. Proportion of catheter-linked complications between inclusion and D16 4.2.2. Number of blood units transfused between inclusion and day 28. 4.2.3. Proportion of major bleeding according to the International Society On Thrombosis And Haemostasis 4.2.4. Proportion of patients with occurrence of an acute renal failure at D28, according to the Kidney Disease Improving Global Outcomes (KDIGO) guidelines 4.2.5. Proportion of patients with anaphylactic reaction at day 28

The experimental design is multicenter, randomized, controlled, open-label superiority trial in parallel groups. The population involved is ICU patients with a Partial pressure of oxygen/ Fraction inspired by oxygen (PaO2/FIO2) ratio < 200 and a diagnosis of acute exacerbation of idiopathic pulmonary fibrosis.

The experimental group will receive a combination of:

1. Methylprednisolone bolus of 1g i.v. day 1, then 20 mg/day (or oral prednisone equivalent) for 21 days;
2. Nine therapeutic plasma exchanges of 1.5x the estimated plasma volumes using albumin:saline (3:1) or fresh frozen plasma in case of an International Normalised Ratio (INR) superior to 1.5, on days 1,2,3,5,7,9,11,13,15; followed by administration of low dose of intravenous immunoglobulin (100 mg/kg)
3. Rituximab 1 g i.v. on days 7 and 15 (after therapeutic plasma exchange and premedication);
4. Intravenous immunoglobulin 0.5 g/kg/d on days 16 to 19.

The reference group will receive:

Intravenous methylprednisolone bolus of 10 mg/kg (max. 1g) on day 1, 2 and 3, then 1 mg/kg/d for 1 week, and 0.75 mg/kg/d for 1 week, then 0.5 mg/kg/d for 1 week, and 0.25 mg/kg/d for 1 week, and 0.125 mg/kg/d until day 90. Shift to oral prednisone as soon as the oral route is available.

Other procedures added by the research:

Blood sampling for serial serum lung injury biomarkers, fibrocytes determination and circulating antibodies measurements

Risks added by the research: C Number of subjects chosen: 40 Number of centres : 17

Research period:

Inclusion period: 36months Length of participation: one year

* Maximum period between selection and inclusion: 3 days
* Treatment period: 90 days
* Follow up period: 1 year +/- 2 weeks
* Total research period: 48 months

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥ 18 years of age
2. Admitted to ICU in the last 72 h
3. Definite or probable IPF diagnosis defined on 2018 ATS/ERS/JRS/ALAT guidelines or a possible usual interstitial pneumonia pattern on HRCT without etiology.
4. Definite AE-IPF according to the 2018 revised criteria :

   1. Previous or concurrent diagnosis of idiopathic pulmonary fibrosis (if the diagnosis of IPF is not previously established, this criterion can be met by the presence of radiologic and or histopathologic changes consistent with usual interstitial pneumonia (UIP) pattern on the current evaluation);
   2. Acute worsening or development of dyspnea typically of less than one-month duration;
   3. Computed tomography with new bilateral ground-glass opacity and/or consolidation superimposed on a background pattern consistent with a UIP pattern (if no previous computed tomography is available, the qualifier "new" can be dropped);
   4. Deterioration not fully explained by cardiac failure or fluid overload.
5. PaO2/FiO2 ratio < 200 measured on FiO2 1

Exclusion Criteria:

1. Known hypersensitivity intravenous immunoglobulins or rituximab
2. Severe heart failure
3. Active and uncontrolled bacterial fungal or parasitic infection ruled out by at least one of these two conditions

   1. Procalcitonin value at inclusion < 0.25 ng/mL OR
   2. Adapted antimicrobial therapy for at least 48 hours at inclusion
4. Positive multiplex PCR for Influenzae A and B, or VRS
5. Deep Veinous Thrombosis or Pulmonary embolism in the last six months
6. Prior exposures to human-murine chimeric antibodies
7. Ongoing treatment with a cellular immunosuppressant (e.g., cyclophosphamide, methotrexate, mycophenolate, azathioprine, calcineurin inhibitors, etc.)
8. Subject treated with more than 2 boluses of methylprednisolone (total dose > 500mg of methylprednisolone) or one dose > 10mg/kg in the last 72 hours
9. Uncorrectable coagulopathies or thrombocytopenia < 30000/mm3
10. Active cancer (other than basal cell carcinoma of the skin)
11. Other source of immunosuppression (i.e. HIV infection, solid organ transplant, lymphoma or leukemia)
12. Pregnancy
13. Patient listed for lung transplantation
14. Patient on ECMO
15. Patient with a do-not-intubate order at inclusion
16. Concurrent participation in other experimental trials
17. Not Affiliation to the French social security
18. Not Written informed consent from the patient or a legal representative if appropriate
19. Hypersensitivity to corticosteroids, cotrimoxazole / atovaquone
20. Patients with severe renal insufficiency (creatine clearance <15ml / min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-05-16 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Overall mortality at day 28 after initiation of therapy (Day1) | 28 days
  Overall mortality at day 28 after initiation of therapy (Day1)

SECONDARY OUTCOMES:
Overall mortality at 12 months | 12 months
  Overall mortality at 12 months
Number of days alive without mechanical ventilation between day 1 and day 28 | 28 days
  Number of days alive without mechanical ventilation
Length of ICU- stay and hospital-stay | 12 months
  Length of ICU- stay and hospital-stay
Evolution of the SOFA score between day 1 and day 28 or discharge-day from ICU as appropriate (in case of death before Day 28, the last SOFA score collected will be 24 points) | 28 days
  The Sequential Organ Failure Assessment (SOFA) score is calculated with the combination of 6 scores:
  * respiratory score with the parameter PaO2/ FiO2
  * neurological score with Mean arterial pressure parameter
  * hepatic score with bilirubin parameter
  * coagulation score with measure of platelets
  * renal score with creatinine parameter
  The total score will range to 0 at 24; 0 being the better outcome and 24 the worse.
Variation of global extent of HRCT infiltrates between initial HRCT and Day 90 according to AKIRA et al | 90 days
  Variation of global extent of HRCT infiltrates
Changes in lung injury biomarkers in plasma (KL-6, SP-D) between day 1 and day 90 | 90 days
  Changes in lung injury biomarkers in plasma
Changes in circulating autoantibodies levels (anti-periplakin, anti-HSP70 and anti-vimentin antibodies) between day 1 and day 90 | 90 days
  Changes in circulating autoantibodies levels
Changes in the proportion of blood fibrocytes between day 1 and day 90 | 90 days
  Changes in the proportion of blood fibrocytes between day 1 and day 90
Proportion of patients with at least one episode of any healthcare-associated infection between inclusion and day 28 | 28 days
  Proportion of patients with at least one episode of any healthcare-associated infection
Proportion of catheter-linked complications between inclusion and day 16 | 16 days
  Proportion of catheter-linked complications between inclusion and day 16
Number of blood units transfused between inclusion and day 28 | 28 days
  Number of blood units transfused between inclusion and day 28
Proportion of major bleeding according to the International Society On Thrombosis and Haemostasis | 28 days
  Proportion of major bleeding
Proportion of patients with occurrence of an acute renal failure at day 28, according to the KDIGO guidelines | 28 days
  Proportion of patients with occurrence of an acute renal failure
Proportion of patients with anaphylactic reaction at day 28 | 28 days
  Proportion of patients with anaphylactic reaction

CONTACTS AND LOCATIONS:
Overall Officials: Bruno CRESTANI, Professor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Bichat Claude Bernard, Paris, France